CLINICAL TRIAL: NCT05256160
Title: Cortical Excitability in Cyclic Vomiting Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, David Levinthal, Assistant Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY21120001
Record Dates: First submitted 2022-02-15; First posted 2022-02-25 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Cyclic Vomiting Syndrome
MeSH Terms: conditions — Familial cyclic vomiting syndrome

STUDY DESIGN:
Intervention Model Description: This is a comparative study looking at differences in electrophysiologic measures of cortical excitability between those with Cyclic Vomiting Syndrome and healthy controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CVS subjects (Experimental): Subjects diagnosed with Cyclic Vomiting Syndrome (CVS)
  Interventions: Other: TMS Paired-Pulse assessment of cortical excitability; Other: Autonomic activity
- healthy, non-CVS subjects (Active Comparator): Subjects not diagnosed with CVS
  Interventions: Other: TMS Paired-Pulse assessment of cortical excitability; Other: Autonomic activity

INTERVENTIONS:
Other: TMS Paired-Pulse assessment of cortical excitability — Using the paired-pulse TMS paradigm, intracortical inhibition and facilitation of cortical circuitry will be assessed by stimulating the motor cortex and using the electromyographic (EMG) response of a target muscle as readout. In such studies, a conditioning stimulus modulates the amplitude of the motor-evoked potential (MEP) produced by the test stimulus. Depending on the inter-stimulus interval, effects can be attributed to different aspects of cortical processing. Brief intervals (1-5 ms) will be used to assess short-interval intracortical inhibition (SICI) and short-interval intracortical facilitation (SICF), intermediate intervals (7-20 ms) to assess intracortical facilitation (ICF) and long intervals (50-200 ms) to assess long-interval intracortical inhibition (LICI).
Other: Autonomic activity — Autonomic function will be determined using continuously recorded EKG and used as covariates to investigate any systematic impact on cortical excitability measures collected with the paired-pulse protocols.

SUMMARY:
This exploratory study will determine if there are differences in cortical excitability between patients suffering from cyclic vomiting syndrome (CVS) and healthy control subjects, as assessed by a non-invasive method of brain stimulation (Transcranial Magnetic Stimulation, TMS).

DETAILED DESCRIPTION:
This exploratory study will determine if there are differences in cortical excitability between patients suffering from cyclic vomiting syndrome (CVS) and healthy control subjects, as assessed by a non-invasive method of brain stimulation (Transcranial Magnetic Stimulation, TMS).

Using the paired-pulse TMS paradigm, intracortical inhibition and facilitation of cortical circuitry will be assessed by stimulating the motor cortex and using the electromyographic (EMG) response of a target muscle as readout. In such studies, a conditioning stimulus modulates the amplitude of the motor-evoked potential (MEP) produced by the test stimulus. Depending on the inter-stimulus interval, effects can be attributed to different aspects of cortical processing. Brief intervals (1-5 ms) will be used to assess short-interval intracortical inhibition (SICI) and short-interval intracortical facilitation (SICF), intermediate intervals (7-20 ms) to assess intracortical facilitation (ICF) and long intervals (50-200 ms) to assess long-interval intracortical inhibition (LICI).

Some clinical, demographic, and autonomic data (i.e. EKG) will be recorded and used as covariates to investigate any systematic impact on cortical excitability measures collected with the paired-pulse protocols.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of CVS

Exclusion Criteria:

* history of CVS (for healthy control population only)
* psychosis or altered cognitive status
* history of head injury, metal in the skull, stroke, or a history of seizures or a history of syncope (fainting or passing out)
* implantable devices, such as a pacemaker or nerve stimulator
* current use of the following medications or use of substances which are known to lower the seizure threshold: clozapine (Clozaril), chlorpromazine (Thorazine), amphetamines or methamphetamine, Ecstasy, Ketamine, Angel Dust/PCP, cocaine, or 3 or more alcoholic drinks per day
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Paired-pulse ratios | Multiple study sessions spanning up to 12 months
  Percentage Change in Paired Pulse (PP) TMS induced MEP responses with inhibitory or facilitatory stimulation.

SECONDARY OUTCOMES:
TMS motor threshold | Multiple study sessions spanning up to 12 months
  TMS stimulator output necessary to elicit 200 microvolt MEP responses
Cortical silent period | Multiple study sessions spanning up to 12 months
  Length (milliseconds) of EMG inactivity following TMS stimulation
Heart rate variability | Multiple study sessions spanning up to 12 months
  Spectral frequency analysis (via Fast Fourier Transformation) of R-R intervals

CONTACTS AND LOCATIONS:
Overall Officials: David J Levinthal, MD PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan to place participant data into a open-access, shared data repository. However, a data sharing agreement can be made if requested.